CLINICAL TRIAL: NCT04936451
Title: Contribution of an Electrotherapy Technique Such as TENS ECOMODYN® vs Electrotherapy Only Type TENS in the Management of Myofascial Syndrome After Breast Surgery
Brief Title: Electrotherapy in the Management of Myofascial Syndrome
Acronym: MODYMYO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recrutment
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: ICO-A-2020-10
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Surgery; Myofascial syndrome
MeSH Terms: conditions — Breast Neoplasms | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Monocentric, randomized in cross over in two arms, open
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS / TENS ECOMODYN (Other): Patients who have signed their consent receive, after randomization, the trial treatments assigned to them. Arm TENS / TENS ECOMODYN Patients first start with TENS during 2 months puis change with TENS ECOMODYN during 2 months with a wash-out period of 15 days
  Interventions: Device: TENS (transcutaneous electrical nerve stimulation); Device: TENS (transcutaneous electrical nerve stimulation) ECOMODYN
- TENS ECOMODYN / TENS (Other): Patients who have signed their consent receive, after randomization, the trial treatments assigned to them. Arm TENS ECOMODYN / TENS Patients first start with TENS ECOMODYN during 2 months puis change with TENS during 2 months with a wash-out period of 15 days
  Interventions: Device: TENS (transcutaneous electrical nerve stimulation); Device: TENS (transcutaneous electrical nerve stimulation) ECOMODYN

INTERVENTIONS:
Device: TENS (transcutaneous electrical nerve stimulation) — Patients will benefit from screening for refractory pain, neuropathic or not, with myofascial syndrome, between 3 and 12 months after surgery.
  The healthcare professional will determine 4 trigger points. TENS is applied twice 45 min every day for 2 months. Pain treatment will be done by using the P6 program in alternative mode: 2hz / 100Hz.
  The time between 2 electrostimulations will be a minimum of 4 hours and a maximum of 15 hours.
Device: TENS (transcutaneous electrical nerve stimulation) ECOMODYN — TENS ECOMODYN® is applied to 4 treatment points, 5 minutes per point 2 times a day for 2 months.
  A minimum rest period of 4 hours between 2 sessions on the same point must be respected Stimulation is performed directly with the bipolar probe of the TENS ECOMODYN® device on the painful area by fixed stimulation of 4 active pain points in 77Hz mode.

SUMMARY:
Myofascial syndrome is defined as "musculoskeletal pain characterized by local and referred pain perceived to be deep and constant, and by the presence of myofascial trigger points in any part of the body" Post-breast surgery myofascial syndrome affects up to 44.7% of operated women, mainly on the muscles of the greater shoulder girdle. The repercussions are significant, functional, somatic, psychological and socio-professional affecting the quality of life. The treatments offered may or may not be medicinal. Transcutaneous electrical nerve stimulation (TENS) is a therapy that uses low voltage electrical current to provide pain relief. A TENS unit consists of a battery-powered device that delivers electrical impulses through electrodes placed on the surface of your skin. The electrodes are placed at or near nerves where the pain is located or at trigger points.

ELIGIBILITY:
Inclusion Criteria:

* Male or female who had first breast cancer surgery, regardless of the type of surgery
* Age ≥ 18 years
* Patients with refractory pain with myofascial syndrome, with a numerical scale ≥ 4
* Topical treatment for refractory pain completed more than 30 days ago
* Healthy, non-irritated skin on painful areas to treat
* Patient with a third party who can attend visits M0 and M2.5
* Obtaining the signed written consent of the patient
* Major patient affiliated to a social security scheme

Exclusion Criteria:

* Patient who has used TENS before on the muscles affected by the myofascial syndrome
* Post-surgery management of the affected area by a physiotherapist
* Person with venous thrombosis
* Contraindications specific to the treatments studied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
The main objective is to evaluate the effectiveness of TENS and TENS ECOMODYN® on the management of chronic breast pain after surgery. | 16,5 months
  Chronic pain is assessed using the Digital Pain Rating Scale (0 worse outcome to 10 better outcome) before and after using the method (TENS and TENS ECOMODYN®) at M0, M2, M2.5 and M4.5.

SECONDARY OUTCOMES:
Evaluate the changes made by the treatment felt by the patient | 16.5 months
  The intensity of The patient's feelings will be evaluated by the Patient Global Impression of Change questionnaire: at M2 and M4.5

CONTACTS AND LOCATIONS:
Overall Officials: EVA KERROUAULT, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (1):
- Institut de Cancerologie de l'Ouest, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: No